CLINICAL TRIAL: NCT01097733
Title: Dual-Source Computed Tomography to Improve Prediction of Response to Cardiac Resynchronization Therapy
Acronym: DIRECT
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Jagmeet Singh, Jagmeet Singh, MD, Massachusetts General Hospital
Other Study IDs: 2008P000555; 1K23HL098370 (NIH)
Record Dates: First submitted 2010-03-25; First posted 2010-04-02 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure - NYHA II - IV; Wide QRS Complex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pre-procedural cardiac CT: CRT patients will undergo pre-procedural cardiac CT to assess for dyssynchrony, scar, and coronary venous anatomy. The CT venogram will be randomize to pre-knowledge to implanting physician or blinded. The CT dyssynchrony and scar assessment will remain blinded to caregivers and patients.
  Interventions: Other: Randomization of Pre-knowledge of CT coronary venography

INTERVENTIONS:
Other: Randomization of Pre-knowledge of CT coronary venography

SUMMARY:
Cardiac Resynchronization Therapy (CRT) is a widely accepted treatment that has led to improved clinical outcomes for patients with refractory congestive heart failure (CHF), systolic dysfunction, and wide QRS duration. However, it requires implantation of an expensive device ($30,000) and about 1/3 of patients do not have clinical improvement. Inadequate amounts of LV dyssynchrony or suboptimal lead placement may limit clinical response. Dual-Source computed tomography (DSCT) allows for subtle detection during myocardial contraction for assessing LV dyssynchrony, and can also assess coronary venous anatomy and scar burden. Thus DSCT may be the ideal noninvasive modality to predict response to CRT.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Ability to provide informed consent
* Planned CRT implantation
* NYHA Functional Class II-IV heart failure
* Echo Ejection Fraction less than or equal to 35%
* QRS duration greater than or equal to 120 ms
* Normal or mildly reduced kidney function (estimated serum creatinine less than or equal to 1.5 mg/dL or less than or equal to 1.3 mg/dL for diabetic subjects on metformin
* For diabetic subjects on glucophage (metformin) they will be required to stop glucophage (metformin) for at least 48 hours after the administration of contrast.

Exclusion Criteria:

* Known allergy to iodine or iodinated contrast
* Chronic persistent atrial fibrillation
* Pregnancy or unknown pregnancy status
* Subjects on glucophage (metformin) therapy that are unable or unwilling to discontinue therapy for 48 hours after CT scan
* Known inadequate venous access for appropriate IV caliber placement
* Iodinated contrast administration within the past 48 hours
* Subjects who cannot hold their breath for 10-15 seconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient or inpatient heart failure patients scheduled for CRT implantation
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Clinical Response to CRT | 6 months post implantation of CRT
  The clinical response to CRT will be adjudicated by two experienced cardiologists taking into account left ventricular ejection fraction, NYHA functional class, and patient global assessment score.

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 2 years
  MACE defined as composite endpoints of death, cardiac transplant, left ventricular assist device, and HF hospitalization
Secondary endpoints | 6 months
  Change in NYHA Functional Class, Echo volumes and ejection fraction, Minnesota Quality of Life score, 6-minute walk distance, NT-proBNP levels, and hospitalization at 6 months

OTHER OUTCOMES:
Implantation and fluoroscopy time and radiation exposure | During time of implant
  Implantation time, fluoroscopy time, and radiation exposure
Agreement between CT venography and invasive coronary venography | within the CT venography and invasive coronary venography

CONTACTS AND LOCATIONS:
Overall Officials: Jagmeet P Singh, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Truong QA, Singh JP, Cannon CP, Sarwar A, Nasir K, Auricchio A, Faletra FF, Sorgente A, Conca C, Moccetti T, Handschumacher M, Brady TJ, Hoffmann U. Quantitative analysis of intraventricular dyssynchrony using wall thickness by multidetector computed tomography. JACC Cardiovasc Imaging. 2008 Nov;1(6):772-81. doi: 10.1016/j.jcmg.2008.07.014. PMID 19212461
- [Derived] Galand V, Ghoshhajra B, Szymonifka J, Das S, Orencole M, Barre V, Martins RP, Leclercq C, Hung J, Truong QA, Singh JP. Left ventricular wall thickness assessed by cardiac computed tomography and cardiac resynchronization therapy outcomes. Europace. 2020 Mar 1;22(3):401-411. doi: 10.1093/europace/euz322. PMID 31865389
- [Derived] Truong QA, Szymonifka J, Picard MH, Thai WE, Wai B, Cheung JW, Heist EK, Hoffmann U, Singh JP. Utility of dual-source computed tomography in cardiac resynchronization therapy-DIRECT study. Heart Rhythm. 2018 Aug;15(8):1206-1213. doi: 10.1016/j.hrthm.2018.03.020. Epub 2018 Mar 20. PMID 29572087